CLINICAL TRIAL: NCT05988710
Title: Low-dose Buccal Buprenorphine: Relative Abuse Potential and Analgesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Daniel Larach, Asst Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 222204; 1K23DA057387 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Analgesia; Abuse Opioids; Pain
MeSH Terms: conditions — Agnosia; Opioid-Related Disorders; Pain

STUDY DESIGN:
Intervention Model Description: randomized, double blind, double-dummy, placebo-controlled, crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Buccal Buprenorphine 300mcg and oral Placebo (Experimental): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Buccal Buprenorphine 300 mcg; Drug: Oral Placebo
- Buccal Buprenorphine 600mcg and oral Placebo (Experimental): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Buccal Buprenorphine 600 mcg; Drug: Oral Placebo
- Buccal Buprenorphine 900mcg and oral Placebo (Experimental): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Buccal Buprenorphine 900 mcg; Drug: Oral Placebo
- Oral immediate release oxycodone 10mg and buccal placebo (Active Comparator): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Buccal Placebo; Drug: Oral immediate-release oxycodone 10mg
- Oral placebo and buccal placebo (Placebo Comparator): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Buccal Placebo; Drug: Oral Placebo
- Buccal Buprenorphine 450mcg and oral Placebo (Experimental): In randomized order (crossover) across 5 laboratory sessions approximately 5 days apart, participants will receive: 1) Buccal buprenorphine 300 mcg and oral placebo, 2) Buccal buprenorphine 450 mcg and oral placebo 3) Buccal buprenorphine 600 mcg and oral placebo, 4) Buccal buprenorphine 900 mg and oral placebo, 5) oral immediate-release oxycodone 10mg and oral placebo, or 6) buccal placebo and oral placebo.
  Interventions: Drug: Oral Placebo; Drug: Buccal Buprenorphine 450mcg

INTERVENTIONS:
Drug: Buccal Buprenorphine 300 mcg — buprenorphine for 300mcg buccal administration
  Arms: Buccal Buprenorphine 300mcg and oral Placebo
Drug: Buccal Buprenorphine 600 mcg — buprenorphine for 600mcg buccal administration
  Arms: Buccal Buprenorphine 600mcg and oral Placebo
Drug: Buccal Buprenorphine 900 mcg — buprenorphine for 900mcg buccal administration. Note: This arm has been discontinued as of 06/25/2024 and has been replaced with the 450mcg buprenorphine buccal administration arm.
  Arms: Buccal Buprenorphine 900mcg and oral Placebo
Drug: Buccal Placebo — Placebo for buccal administration
  Arms: Oral immediate release oxycodone 10mg and buccal placebo; Oral placebo and buccal placebo
Drug: Oral Placebo — Placebo for oral administration
  Arms: Buccal Buprenorphine 300mcg and oral Placebo; Buccal Buprenorphine 450mcg and oral Placebo; Buccal Buprenorphine 600mcg and oral Placebo; Buccal Buprenorphine 900mcg and oral Placebo; Oral placebo and buccal placebo
Drug: Oral immediate-release oxycodone 10mg — Immediate-release oxycodone for 10 mg oral administration
  Arms: Oral immediate release oxycodone 10mg and buccal placebo
Drug: Buccal Buprenorphine 450mcg — buprenorphine for 450mcg buccal administration. Note: This arm has been added to replace the 900mcg buprenorphine buccal administration arm.
  Arms: Buccal Buprenorphine 450mcg and oral Placebo

SUMMARY:
The goal of this study is to compare the abuse potential of low-dose equianalgesic buccal buprenorphine to a commonly used full mu opioid receptor (MOR) agonist in a highly controlled experimental setting. This is a translational study in which healthy participants are phenotyped for psychosocial and Opioid-Use-Disorder-risk-related metrics. In a within-subjects crossover design, 60 participants will receive a standard postoperative oral oxycodone dose (10 mg), placebo, and 3 different doses of buccal buprenorphine across 5 separate sessions. Quantitative Sensory Testing (QST) will be used to evaluate alterations in pain responsiveness relative to placebo across buprenorphine doses and oxycodone, and will compare abuse potential (indexed by the standard FDA drug liking metric) following equianalgesic doses of the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* Intact cognitive status and ability to provide informed consent
* Ability to read and write in English sufficiently to understand and complete study questionnaires
* Age 18-65
* Opioid-naive status (defined as no use of full mu-opioid receptor (MOR) agonist, partial MOR agonist, or mixed agonist/antagonist medications for the prior 3 months by patient report

Exclusion Criteria:

* Liver/kidney disease
* Chronic pain
* Current/prior substance use disorder
* Pregnancy (to avoid fetal drug exposure, with pregnancy tests conducted to confirm eligibility)
* Seizure disorder
* Certain psychiatric conditions (severe depression, bipolar disorder, psychotic disorders)
* Recent use of medications that may interfere with study drug metabolism
* Recent benzodiazepine or opioid use (confirmed via rapid urine screening prior to each lab session)
* The presence of any medical conditions felt by the study physician to render participant unsafe
* Prior allergic reaction or intolerance to oxycodone, buprenorphine, or their analogs (explicitly including moderate-to-severe nausea or vomiting with prior opioids)
* Recent use of marijuana, delta-8 THC, CBD, and similar products
* Recent use of kratom
* Severe asthma
* Long QT syndrome
* Parkinson disease
* Weight <60 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Difference in mean maximum effect score (Emax) of the drug liking visual analog scale (VAS) between oxycodone 10 mg and an equianalgesic dose of buprenorphine | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the drug liking VAS between oxycodone 10 mg and an equianalgesic dose of buprenorphine conditions. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Quantitative sensory testing (QST) thermal pain tolerance in seconds | Baseline through 3.5 hours after study drug administration on each medication condition
  Mean time in seconds elapsed from onset of the heat pain stimulus to participants withdrawal from the stimulus. Heat pain tolerance is an indicator of pain sensitivity. This will determine the equianalgesic dose of buccal buprenorphine compared to oxycodone 10 mg. Equivalence to oxycodone will be defined as the buprenorphine does that produces a mean thermal pain tolerance increase within 0.5 standard deviation of the oxycodone. response.

SECONDARY OUTCOMES:
Difference in mean maximum effect score (Emax) of the drug liking visual analog scale between equianalgesic dose of buprenorphine and placebo conditions | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean maximum effect score (Emax) of the drug liking visual analog scale between equianalgesic dose of buprenorphine and placebo conditions. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
Difference in mean maximum effect score (Emax) of the drug liking visual analog scale between oxycodone 10 mg and placebo conditions | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean maximum effect score (Emax) of the drug liking visual analog scale between oxycodone 10 mg and placebo conditions. Drug liking VAS is a bipolar scale designed to assess a participant's liking for a given study intervention at the time the question is being asked (that is, at this moment). It is scored as an integer ranging from 0 (strong disliking) to 100 (strong liking).
QST heat pain threshold | Baseline through 3.5 hours after study drug administration on each medication condition
  Mean time in seconds elapsed from onset of the thermal stimulus to the point at which heat stimulus is first experienced as painful. Thermal pain threshold is an indicator of pain sensitivity.
Visual Analog Scale (VAS) pain intensity | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the pain intensity VAS between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. The VAS pain intensity is a measure of experienced pain intensity on 0 to 100 scale when 0 is no pain and 100 is worst pain imaginable.
VAS pain unpleasantness | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the pain unpleasantness VAS between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. The VAS pain unpleasantness is a measure of experienced pain unpleasantness on 0 to 100 scale, when 0 is no unpleasantness and 100 is most unpleasant imaginable.
McGill Pain Questionnaire - Short Form | Baseline through 3.5 hours after study drug administration on each medication condition
  Mean of maximum McGill Pain Questionnaire - Short Form score between oxycodone 10mg, equianalgesic dose of buprenorphine and placebo. The score ranges from 0-33 where 0 represents no pain and 33 represents most intense pain. Positive change values indicate decreased pain responsiveness.
VAS alertness/drowsiness | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS alertness/drowsiness between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. The VAS alertness/drowsiness assesses alertness and drowsiness following drug administration on 0 to 100 sale, when 0 is extreme drowsiness, 50 is neutral, and 100 is extreme alertness.
VAS any drug effects | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS any drug effects between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS any drug effects assesses presence of any drug effects felt by participant on 0 to 100 scale, when 0 is no drug effects and 100 is extreme drug effects.
VAS good effects | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS good effects between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS good effects assesses presence of drug effects characterized as good felt by participant on scale 0 to 100 when 0 is no good drug effects and 100 is extreme good drug effects.
VAS feeling high | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS feeling high between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS feeling high assesses presence of "feeling high" by participant on 0 to 100 scale when o is not feeling high at all and 100 is feeling extremely high.
VAS bad effects | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS bad effects between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS bad effects assesses presence of drug effects characterized as bad felt by participant on 0 to 100 scale when 0 is no bad drug effects and 100 is extreme bad drug effects.
VAS desire to use opioids | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS desire to use opioids between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS desire to use opioids assesses participant's desire to use opioids on a 0-100 scale when 0 is no desire to use opioids and 100 is extreme desire to use opioids.
Opioid Adjective Rating Scale | Baseline through 3.5 hours after study drug administration on each medication condition
  Difference in mean Emax of the VAS Opioid Adjective Rating Scale between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo. VAS Opioid Adjective Rating Scale is a 12 item questionnaire which evaluates common sensory and somatic effects of opioid (e.g., itching, vomiting, sweating, nausea, dry mouth). Each effect is rated on 0 to 4 scale when 0 is not at all and 4 is extremely.
Temporal summation of pain (TSP) | Baseline through 3.5 hours after study drug administration on each medication condition
  Change in pain intensity between first and most painful TSP stimuli (mean of two TSP trials) compared between oxycodone 10 mg, equianalgesic dose of buprenorphine and placebo conditions. Pain intensity will be measured on a 0-10 Numeric Rating Scale when when 0 is no pain and 100 is worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Larach, MD, MSTR, MA, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No